CLINICAL TRIAL: NCT04497298
Title: A Randomized, Placebo-controlled Trial, to Evaluate the Safety and Immunogenicity of the COVID-19 Vaccine, a Measles Vector-based Vaccine Candidate Against COVID-19 in Healthy Volunteers Consisting of an Unblinded Dose Escalation and a Blinded Treatment Phase
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of the COVID-19 Vaccine
Acronym: COVID-19-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Themis Bioscience GmbH (Industry); Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-016; 2020-002973-89 (EudraCT Number)
Record Dates: First submitted 2020-07-31; First posted 2020-08-04 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-07

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Vaccine; Prevention
MeSH Terms: conditions — COVID-19 | interventions — Organization and Administration

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As safety precaution, the study will begin with enrollment of two successive unblinded dose groups of sentinel participants randomized into groups of three in an open-label fashion (group A and B). All site personnel, Sponsor and participants will be unblinded.
  Then remaining participants will be randomized in a blinded manner to one of three cohorts (A, B, C) and between vacccine candidate and placebo. Site personnel responsible for study medication handling, preparation and Administration will be unblinded, only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COVID-19 vaccine candidate (TMV-083/V-591) - Low dose (Experimental): Volunteers will receive two administrations of the low dose COVID-19 vaccine candidate by intramuscular (i.m.) injection on day 0 and 28
  Interventions: Biological: Two COVID-19 vaccine candidate (TMV-083/V-591) administrations - Low dose
- COVID-19 vaccine candidate (TMV-083/V-591) - High dose (Experimental): Volunteers will receive two administrations of the high dose COVID-19 vaccine candidate by intramuscular (i.m.) injection on day 0 and 28.
  Interventions: Biological: Two COVID-19 vaccine candidate (TMV-083/V-591) administrations - High dose
- One COVID-19 vaccine candidate (TMV-083/V-591) - High and placebo (Experimental): Volunteers will receive one administration of the high dose COVID-19 vaccine candidate on day 0 by intramuscular (i.m.) injection and one administration of the placebo on day 28 by intramuscular (i.m.) injection.
  Interventions: Biological: One COVID-19 vaccine candidate (TMV-083/V-591) administration - High dose; Other: Placebo
- Placebo (Placebo Comparator): Volunteers will receive physiological saline solution (0.9% NaCl), administered by intra muscular (i.m.) injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Two COVID-19 vaccine candidate (TMV-083/V-591) administrations - Low dose — Live-attenuated recombinant measles vaccine virus vector expressing a modified surface glycoprotein of the novel Coronavirus (SARS-CoV-2)
  Arms: COVID-19 vaccine candidate (TMV-083/V-591) - Low dose
Biological: Two COVID-19 vaccine candidate (TMV-083/V-591) administrations - High dose — Live-attenuated recombinant measles vaccine virus vector expressing a modified surface glycoprotein of the novel Coronavirus (SARS-CoV-2)
  Arms: COVID-19 vaccine candidate (TMV-083/V-591) - High dose
Biological: One COVID-19 vaccine candidate (TMV-083/V-591) administration - High dose — Live-attenuated recombinant measles vaccine virus vector expressing a modified surface glycoprotein of the novel Coronavirus (SARS-CoV-2) and placebo
  Arms: One COVID-19 vaccine candidate (TMV-083/V-591) - High and placebo
Other: Placebo — Physiological saline solution (0.9% NaCl)
  Arms: One COVID-19 vaccine candidate (TMV-083/V-591) - High and placebo; Placebo

SUMMARY:
This is a randomized, placebo-controlled, two center, Phase I trial in healthy adult volunteer participants consisting of two phases, an unblinded dose escalation and a double blind treatment phase to investigate the safety, tolerability and immunogenicity of a novel measles-vector based vaccine candidate against SARS-CoV-2 infection (TMV-083/V-591).

DETAILED DESCRIPTION:
This is a prospective, interventional, randomized, Phase I trial comparing two different dose levels and immunization regimen of a novel COVID-19 vaccine candidate (TMV-083/V-591) against SARS-CoV-2 infection, consisting of two phases, an unblinded dose escalation and a double-blind treatment phase, to assess the safety, tolerability and immunogenicity.

90 subjects will be enrolled, 30 per cohort in three cohorts, each cohort comprising 24 vaccinees and 6 placebo recipients. Subjects will either receive two immunizations with a low dosage vaccine (Cohort A), two immunization with a high dosage vaccine (Cohort B), a single immunization with the high dosage vaccine (Cohort C) or placebo (randomized to all three cohorts).

As safety precaution, the study will begin with the enrolment of a small group of 6 sentinel subjects (2 Sentinel Groups, three subjects each of cohorts A and B) each of whom will receive the vaccine on days 0 and 28 in an unblinded and non-randomized manner.

Thereafter, 84 remaining participants will be enrolled in a double-blinded, randomized manner into one of the three cohorts (A, B or C). Placebo will be applied to blind the different regimen.

After the screening visit, participants will be expected to return to the investigational clinical site for 8 visits (9 for the sentinel groups) up to day 91 for immunogenicity sample collection and up to day 210 for safety assessments.

Samples for measles shedding will be collected from subjects of the Sentinel Groups (unblinded regiment in cohort A and B). Body fluids including saliva, nasal swab, urine and whole blood will be collected from day 0 up to day 42.

The investigator and site personnel assessing Adverse Events (AEs), all participants, as well as the sponsor's representatives involved in the monitoring and conduct of the study will be unblinded to which vaccine was administered within the unblinded treatment phase. Only the site personnel performing randomization, preparation and administration of Investigational Medicinal Product (IMP) will be unblinded within the randomized double-blinded treatment phase.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18 and 55 years (at the time of consent).
2. Healthy participant, according to the investigator's clinical judgment, as established by medical history, vital signs, physical examination, and laboratory assessments
3. Participant with a body mass index (BMI) <30.0 kg/m2
4. Provide written informed consent before initiation of any study procedures.
5. A female participant is eligible for this study if she is not pregnant, given by a negative serum pregnancy test at screening and a negative urine pregnancy test at V1 (1st injection), or breast feeding and 1 of the following:

   * Of non-childbearing potential (i.e., women who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses in greater than or equal to 1 year).
   * Of childbearing potential but has been and agrees to continue practicing highly effective contraception or abstinence (if this is the preferred and usual lifestyle of the participant) from 30 days prior to vaccination up to 6 months after the last injection (D210).
   * Highly effective methods of contraception include 1 or more of the following:

     * male partner who is sterile (vasectomised) prior to the female participants entry into the study and is the sole sexual partner for the female participant;
     * hormonal (oral, intravaginal, transdermal, implantable or injectable);
     * an intrauterine hormone-releasing system (IUS);
     * an intrauterine device (IUD) with a documented failure rate of < 1%.
6. A female participant is eligible if she is willing to abstain from donating oocyte from the screening visit up to 6 months after the last injection (D210);
7. A male participant who is sexually active is eligible if he is willing to :

   * use a condom (with/without spermicidal product) from the screening visit up to 6 months after the last injection (D210) except if the male participant is sterile (e.g. vasectomised); the unique female sexual partner is postmenopausal (defined as no menses for 12 months without an alternative medical cause), is permanently sterilized (e.g. hysterectomy or tubal ligation), or use a highly effective methods of contraception;
   * not donate sperm from the screening visit up to 6 months after the last injection (D210);
   * not plan to father a child from the screening visit up to 6 months after the last injection (D210).
8. Negative HIV 1/2 antibody/antigen test, Hepatitis B surface antigen (HBsAg), and Hepatitis C virus (HCV) antibody.
9. Able to understand and comply with planned study procedures and willing to be available for all study-required procedures, visits and calls for the duration of the study.
10. Willing to abstain from donating whole blood or blood derivatives, tissue or organ all along the study.
11. Affiliated to a social security system, (except state medical aid) (Only for France).
12. Volunteer registered in the French Health Ministry computerized file and authorized to participate in a clinical trial (only for France).

Exclusion Criteria:

1. Subjects actively or previously infected by SARS-CoV-2, as determined by a positive RT-PCR and positive serology test.
2. Subject currently working with high risk of exposure to SARS-CoV-2 (e.g. health care worker, emergency response personnel, etc.) or considered at the investigator's discretion to be at increased risk to acquire SARS-CoV-2 for any other reason.
3. Previous vaccination with an investigational COVID-19 vaccine.
4. History of presence of pulmonary disorders (e.g. COPD, etc.) or asthma.
5. History or present of thrombocytopenia and/or bleeding disorders.
6. A positive serum pregnancy test at screening or urine pregnancy test prior to study injection, women who are planning to become pregnant during the study, or women who are breastfeeding.
7. Clinically relevant history of or current renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, hematological, endocrine, inflammatory, autoimmune, central nervous system or neurological diseases or clinically relevant abnormal laboratory values.
8. Use of immunosuppressive drugs like e.g. corticosteroids (excluding topical preparations and inhalers) within 3 months prior to the first vaccination or 6 months for chemotherapies and all along the study.
9. A diagnosis of schizophrenia, bipolar disease, or history of hospitalization for a psychiatric condition or previous suicide attempt.
10. A history of treatment for any other psychiatric disorder in the past 3 years that increases the risk to the subject in the opinion of the investigator.
11. Received immunoglobulin or other blood product within 3 months prior to enrollment or planned receipt of immunoglobulin or a blood product through study completion.
12. Vaccination within 4 weeks prior to first injection or planning to receive a licensed vaccine before D56 (e.g. Inactivated influenza vaccine).
13. Received measles-containing vaccine within 3 months prior to enrollment.
14. History of severe adverse reactions to vaccine administration, including anaphylaxis and related symptoms, such as urticaria, respiratory difficulty, angioedema and abdominal pain to vaccines, or history of known or suspected allergic reaction likely to be exacerbated by any component of the COVID-19 vaccine.
15. Participation in another investigational clinical study within four weeks before the screening visit or planned before the study completion.
16. Individuals who are living and/or working with severely immunocompromised people, pregnant women, lactating women, children under 12 months old, or any other individual that, in the judgment of the investigator, might be at increased risk.
17. Any condition that, in the opinion of the investigator, may interfere with the aim of the study or the safety or wellbeing of the subject.
18. Subjects with any condition associated with, or that might be associated with, an increased risk of severe illness from COVID-19 according to US CDC definition .
19. Subjects with confirmed or suspected immunodeficiency.
20. Exposure to an individual with confirmed COVID-19 or SARS-CoV-2 infection within the past 2 weeks prior to enrollment.
21. Subject with an acute disease and/or fever (body temperature ≥ 38°C) at the time of the 1st vaccination visit.
22. History of confirmed SARS-CoV or MERS-CoV infection.
23. Current heavy smoker defined as smoking at least 20 cigarettes (1 pack, or equivalent) per day or former heavy smoker who was an active heavy smoker within the last year prior to the screening visit or has a total smoking history of ≥ 1 pack per day for 10 years or more.
24. Current or history of alcohol or drug abuse during the previous 3 years.
25. Presence of tattoos that, in the opinion of the investigator, would preclude evaluation of the injection site.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of the COVID-19 vaccine following one or two consecutive intramuscular injections in healthy volunteers | up to Day 210
  Rate of solicited Adverse Event up to 14 days after each injection. Rate of unsolicited AE up to 28 days after the last injection. Rate of serious adverse events (SAEs), serious adverse reactions (SARs), suspected unexpected serious adverse reactions (SUSARs) and adverse events of special interest (AESI) all along the study period (up to Day 210).

SECONDARY OUTCOMES:
To assess induction of SARS-CoV-2 spike protein-binding antibodies upon one or two administrations of the COVID-19 vaccine by means of ELISA up to study day 56 | Day 56
  SARS-CoV-2 specific antibodies up to study day 56 as measured by spike protein-specific ELISA and serum neutralization assay
To assess induction of SARS-CoV-2 neutralizing antibodies upon one or two administrations of the COVID-19 vaccine by means of serum neutralization assay up to study day 91 | Day 91
  SARS-CoV-2 specific antibodies up to study day 91 for each cohort as measured by spike protein-specific ELISA and serum neutralization assay
To assess SARS-CoV-2 spike protein-specific, cell-mediated immune responses up to study day 91, induced by one or two doses of vaccine, by means of intracellular staining and flow cytometry. | up to Day 91
  SARS-CoV-2 spike protein-specific cell-mediated immune response up to study day 91 induced by one or two doses as measured by intracellular staining and flow cytometry
To assess potential measles virus shedding by means of RT-qPCR of saliva, nasal swab, urine, or blood samples in sentinel groups on day 0 and up to day 42 | up to Day 42
  Occurrence of measles virus shedding as evidenced by a positive RT-PCR for saliva, nasal swab, urine, or blood sample in sentinel groups.

OTHER OUTCOMES:
To assess the anti-measles antibody levels at baseline and on day 28 and on day 56 by ELISA | up to Day 56
  Measles virus antibody levels as assessed by standard ELISA assays on day 0 and day 28, and day 56
To assess the natural exposure of the subjects to SARS-CoV-2 during the duration of the trial by means of N protein-specific ELISA | Day 91
  SARS-CoV-2 N protein specific antibody up to study day 91 as measured by immunoassay to differentiate the response to the COVID-19 vaccine from infection
To assess the occurrence of COVID-19 cases in study participants all along the duration of the study | Day 210
  Occurrence of confirmed COVID-19 (i.e. asymptomatic, paucisymptomatic or symptomatic) cases in the study participant all along the study period

CONTACTS AND LOCATIONS:
Overall Officials: Christiane GERKE, PhD, Study Director — Institut Pasteur; Odile LAUNAY, MD, PhD, Principal Investigator — CIC 1417 Cochin-Pasteur
Locations (2):
- SGS Life Sciences, Clinical Pharmacology Unit, Antwerp, Belgium
- CIC Cochin - Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Launay O, Artaud C, Lachatre M, Ait-Ahmed M, Klein J, Luong Nguyen LB, Durier C, Jansen B, Tomberger Y, Jolly N, Grossmann A, Tabbal H, Brunet J, Gransagne M, Choucha Z, Batalie D, Delgado A, Mullner M, Tschismarov R, Berghmans PJ, Martin A, Ramsauer K, Escriou N, Gerke C. Safety and immunogenicity of a measles-vectored SARS-CoV-2 vaccine candidate, V591 / TMV-083, in healthy adults: results of a randomized, placebo-controlled Phase I study. EBioMedicine. 2022 Jan;75:103810. doi: 10.1016/j.ebiom.2021.103810. Epub 2022 Jan 16. PMID 35045362